CLINICAL TRIAL: NCT04722185
Title: Evaluation of the Veriton SPECT/CT System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Carrie Hruska, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-001511
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Focus of Study is Comparison of 2 Types of Gamma Cameras

STUDY DESIGN:
Intervention Model Description: each patient will have 2 scans - one on a conventional system and one on the newer technology
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Evaluation of the Veriton SPECT/CT system (Experimental): To determine if the Veriton system can achieve equal or better image quality than a standard SPECT/CT system.
  Interventions: Diagnostic Test: Veriton SPECT/CT

INTERVENTIONS:
Diagnostic Test: Veriton SPECT/CT — The Veriton system represents an FDA approved (510k cleared) new generation of SPECT/CT systems. It consists of 12 small gamma cameras arrayed in a circle around the patient, and is coupled to a 64-slice CT system.

SUMMARY:
The main purpose of this study is to evaluate a new type of gamma camera (the Veriton system) that provides a significant gain in system sensitivity and improved image quality compared to a conventional gamma camera that can achieve equal or better image quality than a standard SPECT/CT system.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 years or older.
* Currently scheduled to undergo a nuclear medicine exam.

Exclusion Criteria:

* Individuals under 18 years of age.
* Unwilling/unable to sign an informed consent form.
* Unable to lie on a Veriton imaging table for up to 40 minutes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Image quality | 1 year
  Assessment of relative image quality between the Veriton system and a conventional gamma camera as a function of the type of nuclear medicine exam.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Hruska, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States